CLINICAL TRIAL: NCT05674227
Title: Cost-effectiveness Evaluation of Robotic Surgery, Compared to Thoracoscopic and Open Surgery, in the Removal of Lung Lesions Based on "Real-world" Efficacy and Cost Data From the ATS of Milan
Brief Title: Cost-effectiveness Evaluation of Robotic Surgery in the Removal of Lung Lesions in the ATS of Milan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Agenzia di Tutela della Salute della Città Metropolitana di Milano (Other Government)
Collaborators: Istituto Europeo di Oncologia (Other); Humanitas Hospital, Italy (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Ospedale San Raffaele (Other); ASST Grande Ospedale Metropolitano Niguarda (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); ASST Ovest Milanese, Ospedale Nuovo di Legnano (Unknown); IRCCS Multimedica (Other)
Responsible Party: Sponsor
Other Study IDs: 2699
Record Dates: First submitted 2022-12-02; First posted 2023-01-06 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer
Keywords: Robotic surgery; Cost-effectiveness evaluation; Real-world data
MeSH Terms: conditions — Lung Neoplasms | interventions — Robotic Surgical Procedures; Thoracic Surgery, Video-Assisted; Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic surgery: Patients who have undergone pulmonary robotic surgery
  Interventions: Procedure: Robotic surgery
- VAT surgery: Patients who have undergone pulmonary video-assisted thoracoscopy surgery (VATS)
  Interventions: Procedure: Video-assisted thoracoscopy
- Open surgery: Patients who have undergone pulmonary open surgery
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Robotic surgery — Surgical treatment of operable lung cancers using robotic systems
  Groups: Robotic surgery
Procedure: Video-assisted thoracoscopy — Surgical treatment of operable lung cancers using a video-assisted thoracoscopy approach (VAT)
  Groups: VAT surgery
Procedure: Open surgery — Surgical treatment of operable lung cancers using open surgery
  Groups: Open surgery

SUMMARY:
The goal of this observational study is to compare cost-effectiveness of robotic surgery with open surgery and video-assisted thoracoscopy surgery (VATS) in adult patients, resident in the ATS of Milan area, operated for lung cancer.

The main question it aims to answer is:

• Is the robotic surgery cost-effective compared with thoracotomy and VATS in the surgical treatment of operable lung cancers in the adult population of the ATS of Milan?

Researchers will compare robotic surgery with open and VAT surgery of operable lung cancer to see if robotic surgery performs better in terms of cost per year of life gained or in terms of cost per quality of life earned.

DETAILED DESCRIPTION:
Single multicenter retrospective observational study with Real World Evidence (RWE) approach, i.e. an evaluation that uses real-world data (RWD) derived from healthcare flows of the ATS of Milan and data provided by participating centers on the basis of medical records/ clinical databases, both as regards the analysis of efficacy and safety and as regards the economic evaluation of direct costs.

For the analysis of quality of life and the calculation of QALYs (quality-adjusted life years), validated questionnaires will be prospectively administered to the participating subjects. The Epidemiology Unit of the ATS of Milan is the study promoter and it will coordinate the collection of data and will carry out the statistical and economic analyses. Other participating centers will be the thoracic surgeries of the ATS hospitals, which carried out in 2019 (last pre-pandemic COVID-19 year) at least 50 lung operations.

As for the retrospective part of the study, both for the evaluation of clinical efficacy and of costs, the investigators will include all adult subjects (age equal or over 18 years of age at the time of surgery) residents in the ATS of Milan, who were hospitalized between 01/01/2016 and 31/12/2021 for pulmonary surgery (operation codes in any position of the hospital discharge summary form (SDO-Scheda di Dimissione Ospedaliera) and whose hospitalization is present in the SDO database of the ATS of Milan in one of the participating centers. For the evaluation of cost-effectiveness in malignant tumors, subjects with metastases at diagnosis will be excluded.

As for the prospective part of the study, all subjects who will undergo lung surgery during 2023 at the participating centers and will give their consent to participate in the study by signing the informed consent form at the pre-hospitalization or at hospitalization before surgery will be eligible to be enrolled. To evaluate the quality of life PROMs related, the investigators will use the generic questionnaire EuroQol-5 Dimension (EQ-5D-5L) and the specific European Organization for Researchand Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORCT QLQ-LC29), which are available and validated in Italian. The pre-intervention questionnaire will be completed on paper during hospitalization before the intervention or at pre-admission and the data will be entered into the web application of the ATS of Milan by dedicated staff. The subsequent questionnaires at day 7 and 30 can be self-completed by patients or electronically, using the dedicated web application of the ATS of Milan or in paper form, by filling in the documents issued on discharge for this purpose

The cost-effectiveness evaluation will be conducted according to the CHEERS (Consolidated Health Economic Evaluation Reporting Standards) guidelines.

ELIGIBILITY:
Inclusion Criteria:

Retrospective study

* Patients operated on for a lung tumor in the participating Centers from 01/01/2016 to 12/31/2021
* Residents in the ATS of Milan area
* Hospitalization is present in the hospital discharge summary form database of the ATS of Milan

Prospective study

* Patients operated on for lung tumor in the participating Centers from 01/01/2023 to 06/30/2023, who give their consent to be enrolled in the study
* Residents in the ATS of Milan area

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective study will include all adult subjects (age equal or over 18 years of age at the time of surgery) residents in the ATS of Milan, who were hospitalized between 01/01/2016 and 31/12/2021 for pulmonary surgery and whose hospitalization is present in the hospital discharge summary form database of the ATS of Milan in one of the participating centers. For the evaluation of cost-effectiveness in malignant tumors, subjects with metastases at diagnosis will be excluded.
  As for the prospective part of the study, all subjects who will undergo lung surgery during the first six month of 2023 at the participating centers and will give their consent to participate in the study by signing the informed consent form at the pre-hospitalization or at hospitalization before surgery will be eligible to be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-effectiveness ratio (ICER) of robotic surgery for the treatment of operable lung cancer | The time horizon of the evaluation will be limited to 5 years from the intervention and the purchase of the technology.
  The ICER of robotic surgery compared with both VATS and open surgery is defined as the ratio between incremental costs associated with robotic surgery and the variation in effectiveness. Costs will be measured in Euros. Effectiveness will be considered both in terms of life years gained, measured in years, and in terms of quality of life gained, measured in QALY. In the first case, ICER will be measured as Euros/years; in the second, it will be measured as Euros/QALY. It will be evaluated in the treatment of operable lung cancer.

SECONDARY OUTCOMES:
Incremental Cost-effectiveness ratio (ICER) of robotic surgery for the treatment of benign lung lesions | The time horizon of the evaluation will be limited to 5 years from the intervention and the purchase of the technology.
  The ICER of robotic surgery compared with both VATS and open surgery will be evaluated in the treatment of benign lesions in the same population considered for the primary outcome. ICER is defined as the ratio between incremental costs associated with robotic surgery and the variation in effectiveness. Costs will be measured in Euros. Effectiveness will be considered both in terms of life years gained, measured in years, and in terms of quality of life gained, measured in QALY. In the first case, ICER will be measured as Euros/years; in the second, it will be measured as Euros/QALY.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT05674227/Prot_SAP_000.pdf